CLINICAL TRIAL: NCT03251573
Title: The Cohort Study of Cognitive Impairment and Its Association With Clinical Outcomes in Chinese Maintenance Hemodialysis Patients
Brief Title: The Cohort Study of Cognitive Impairment in Chinese Hemodialysis Patients
Acronym: CODE
Status: Completed | Type: Observational
Sponsor: Beijing Shijitan Hospital, Capital Medical University (Other)
Responsible Party: Principal Investigator, Yang Luo, Chief, MD, PhD, Director of nephrology, Beijing Shijitan Hospital, Capital Medical University
Other Study IDs: Z161100002616005
Record Dates: First submitted 2017-08-14; First posted 2017-08-16 (Actual); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Cognitive Impairment; Hemodialysis Complication; Outcome; Neuropsychological Tests
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normal cognitive function: The cognitive impairment classification algorithm We classified subjects as having no, mild, or major cognitive impairment using criteria from the fifth version of the Diagnostic and Statistical Manual of Mental Disorders (DSM-V) as a guideline.20 The age and/or education-adjusted raw score of each individual cognitive test was calculated and compared with the age and/or education-adjusted published norms for Chinese populations.14 Specifically, age- and education-adjusted scores less than 1.5 standard deviations (SDs) below the adjusted mean of the published population norms on all tests in all domains indicated no cognitive impairment; scores of 1.50 to 1.99 SDs and 2.0 or more SDs below the adjusted mean of the published norms on at least one test in at least one domain indicated mild cognitive impairment and major cognitive impairment, respectively
- cognitive impairment: The cognitive impairment classification algorithm We classified subjects as having no, mild, or major cognitive impairment using criteria from the fifth version of the Diagnostic and Statistical Manual of Mental Disorders (DSM-V) as a guideline.20 The age and/or education-adjusted raw score of each individual cognitive test was calculated and compared with the age and/or education-adjusted published norms for Chinese populations.14 Specifically, age- and education-adjusted scores less than 1.5 standard deviations (SDs) below the adjusted mean of the published population norms on all tests in all domains indicated no cognitive impairment; scores of 1.50 to 1.99 SDs and 2.0 or more SDs below the adjusted mean of the published norms on at least one test in at least one domain indicated mild cognitive impairment and major cognitive impairment, respectively
  Interventions: Other: cognitive impairment

INTERVENTIONS:
Other: cognitive impairment — one are of patients were exposed to cognitive impairment
  Groups: cognitive impairment

SUMMARY:
This study is going to apply neuropsychological battery tests to measure cognitive function across multiple cognitive domains in our cohort of 600 maintenance hemodialysis patients and evaluate:

1. The presence and patterns of cognitive impairment in domains of executive function, perceptual-motor function, language, learning and memory, and complex attention;
2. Clinical characteristics of participants with and without cognitive impairment;
3. the risk factors which might be related to cognitive impairment in this group of population;
4. The association between cognitive impairment and all-cause mortality, stroke and non-fatal cardiovascular events;

We hypothesize that hemodialysis patient is going to have cognitive impairment which might be associated with some risk factors. We also anticipate that cognitive impairment might have some kind of association with the clinical outcomes like all-cause mortality, stroke and other common clinical outcomes that we mentioned above.

DETAILED DESCRIPTION:
Neuropsychological assessment All neuropsychological assessments were performed by the research staff that was centrally trained and certified by the study neuropsychologist to conduct the assessments before study commencement. All research staff and patients were native Chinese speakers. Neuropsychological assessment was conducted individually in a separate room on the day after a dialysis session and required on average approximately 90 minutes. Global cognitive function was screened by the Chinese Beijing version of the Montreal Cognitive Assessment (MoCA-BJ).10 The comprehensive battery of neuropsychological tests was designed to assess five cognitive domains: (1) attention/processing speed, using Symbol Digit Modalities Test and the Chinese modified version of the Trail Making Test A,11,12(2) executive function, using the Chinese modified version of the Trail Making Tests B , and a modified version of the Stroop Color-Word Test;13 (3) verbal memory, using the Chinese version of the Auditory Verbal Learning Test for short-delay and long-delay free recall14 and Complex Figure for visual memory (delayed recall test; Chinese version);12 (4) language, using the Chinese modified versions of Boston Naming Test (the 30-item version) and Animal Fluency Test;15,16and (5) visuospatial function, using the Rey-Osterrieth Complex Figure (copy test).17,18 Depression was assessed using the Hamilton Depression Scale, with scores ranging from 0 to 63 and a score of 7 or above suggested as the optimal cutoff for suspected depression.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects have end-stage kidney disease and are treated with long-term outpatient haemodialysis in each investigational site for at least the previous 3 months;
2. 50 ~ 80 years old;
3. willing to provide written and informed consent.

Exclusion Criteria:

1. Subjects have disturbance of consciousness or mental disorder;
2. Subjects have sensory (visual and hearing) or motor impairment, which disabled them to complete the tests that required these senses;
3. Subjects have a life expectancy less than 6 months according to their physician, have a planned kidney transplantation within 6 months of baseline, or have anticipated recovery of kidney function.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese Maintenace Hemodialysis Patients
Sampling Method: Non-Probability Sample
Enrollment: 613 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-06-18 (Actual); Study Completion 2019-06-18 (Actual)

PRIMARY OUTCOMES:
cognitive function | This measurement is going to be completed within 3 months after the first participant enrolls.
  This study is going to apply neuropsychological battery tests to measure cognitive function across multiple cognitive domains

CONTACTS AND LOCATIONS:
Overall Officials: Yang Luo, MD, PhD, Principal Investigator — Beijing Shijitan Hospital Affiliated to Capital Medical University
Locations (1):
- Beijing Shijitan Hospital affiliated to Capital Medical University, Beijing, China

REFERENCES:
- [Derived] Tian R, Bai Y, Guo Y, Ye P, Luo Y. Association Between Sleep Disorders and Cognitive Impairment in Middle Age and Older Adult Hemodialysis Patients: A Cross-Sectional Study. Front Aging Neurosci. 2021 Dec 8;13:757453. doi: 10.3389/fnagi.2021.757453. eCollection 2021. PMID 34955811